CLINICAL TRIAL: NCT07079475
Title: A Phase I/II, Open-Label, Multicenter Study to Assess the Safety, Tolerability, Pharmacokinetics, and Anti-tumor Efficacy of DZD6008 Combined With Sunvozertinib in Patients With Advanced Non-small Cell Lung Cancer (NSCLC) With EGFR Mutations (TIAN-SHAN8)
Brief Title: Study of Oral EGFR Inhibitor DZD6008 Combined With Sunvozertinib in Patients Who Have Advanced NSCLC With EGFR Mutations (TIAN-SHAN8)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dizal (Jiangsu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Dizal Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DZ2025C0001
Record Dates: First submitted 2025-07-10; First posted 2025-07-23 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DZD6008 + Sunvozertinib (Experimental)
  Interventions: Drug: DZD6008; Drug: Sunvozertinib
- Osimertinib (Active Comparator)
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: DZD6008 — DZD6008 will be administered orally at 40/60 mg QD or selected dose.
  Arms: DZD6008 + Sunvozertinib
Drug: Sunvozertinib — Sunvozertinib will be administered orally at 100 mg QD or selected dose.
  Arms: DZD6008 + Sunvozertinib
Drug: Osimertinib — Osimertinib will be administered orally at 80 mg QD
  Arms: Osimertinib

SUMMARY:
This study will treat patients with advanced NSCLC harboring EGFR mutations. This is the first study to test DZD6008 combined with sunvozertinib in patients, which will help to understand what type of side effects with the treatment. It will also measure the levels of two drugs in the body and preliminarily assess the anti-tumor activity with the combination treatment

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be able to provide documented informed consent.
2. Aged ≥ 18 years.
3. Histologically or cytologically confirmed diagnosis of non-squamous NSCLC, locally advanced or metastatic, not suitable for curative therapy.
4. Documentation of EGFR mutation from a local certified laboratory. Part A: EGFR mutations (excluding participants only harboring EGFR exon20ins). Part B: EGFR sensitizing mutations (Exon19del and/or L858R) with or without T790M/C797S resistance mutations.
5. Provide adequate baseline tumor and plasma samples. For part A: tumor samples collected after disease progression on the last EGFR TKI treatment. For part B: tumor samples of B1 and B2 cohorts should be collected after disease progression on the last EGFR TKI treatment. Tumor samples of B3 cohort should be collected before the study treatment.
6. Previous anti-tumor therapy requirement. For part A, B1, and B2 cohorts of part B: participants should have failed (progressed on or are intolerant to) one line of third-generation EGFR TKI regimen (such as Osimertinib), with (cohort B2) or without (cohort B1) prior platinum-based chemotherapy treatment. Participants could receive no more than 2 lines of EGFR TKI treatment and no more than 3 lines of systemic therapy. Participants in B3 cohort: should not receive prior systemic anti-tumor therapy.
7. ECOG 0 or 1 with predicted life expectancy ≥ 12 weeks.
8. Brain metastases must be stable at study entry.
9. Measurable disease per RECIST 1.1.
10. Adequate hematopoietic and other organ system functions.

Exclusion Criteria:

1. NSCLC with mixed small-cell lung cancer (SCLC) or NSCLC with histologic SCLC transformation.
2. For part A: participants only harboring EGFR exon20ins（harboring other EGFR mutations could be enrolled）.
3. Prior treatment with any of the following: 1) Previously received two or more than two lines of third-generation EGFR TKI treatment. 2) Previously received systemic anti-cancer therapy for advanced disease (only for B3 cohort). 3) Immunotherapy or other antibody therapy within 4 weeks prior to the first administration; 4) Any cytotoxic chemotherapy, investigational drugs or other anticancer drugs from a previous treatment regimen or clinical study within 14 days prior to the first administration; 5) Radiotherapy with a limited field of radiation for palliation within 7 days of the first administration, radiation to more than 30% of the bone marrow or with a wide field of radiation within 28 days of the first administration; 6) Currently receiving or unable to stop drug or herbal supplements known to be potent inhibitors or inducers of cytochrome P450 (CYP)3A4. A washout period of at least 2 weeks for strong inhibitors and 3 weeks for strong inducers is required prior to the first study drug administration; 7) Currently receiving or unable to stop drugs known to be CYP3A4 sensitive substrate with a narrow therapeutic index. A washout period of at least 2 weeks is required prior to the first study drug administration; 8) Currently receiving or unable to stop drugs known to be proton-pump inhibitors. A washout period of at least 1 week is required prior to the first study drug administration; 9) Major surgery within 4 weeks of the first administration of study drug administration or anticipated during the study period.
4. Any unresolved toxicities from prior anti-cancer therapy greater than CTCAE Grade 1.
5. Spinal cord compression or leptomeningeal metastasis.
6. Participants with any other malignancy within 2 years of the first administration of the study drug.
7. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses as judged by the investigator.
8. Participants with active infection, including but not limited to HBV, HCV and HIV.
9. Resting QTcF > 470 msec; Any clinically significant abnormalities in rhythm, conduction or morphology of resting ECG; Any factors that increase the risk of QTc prolongation.
10. Past medical history of ILD or active ILD.
11. Diseases that would preclude adequate absorption of study drug.
12. Received a live vaccine within 2 weeks before the first administration of study drug.
13. Women who are pregnant or breastfeeding.
14. Hypersensitivity to active or inactive excipients of DZD6008, sunvozertinib or osimertinib (only for B3 cohort).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Part A: To assess safety and tolerability | Through the study completion, an average of around 2 years
  Number of participants with Adverse events (AEs)/Serious adverse events (SAEs)
Part A: To assess safety and tolerability | 21 days after the first dose
  Number of participants with Dose-limiting Toxicities (DLTs)
Part B: To assess anti-tumor activity | Through the study completion, an average of around 2 years
  Objective Response Rate (ORR) assessed by investigator per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

SECONDARY OUTCOMES:
Part A: To assess the anti-tumor activity | Through the study completion, an average of around 2 years
  ORR assessed by investigator per RECIST version 1.1
Part A: To assess the anti-tumor activity | Through the study completion, an average of around 2 years
  Duration of Response (DoR) assessed by investigator per RECIST version 1.1
Part A: To assess the anti-tumor activity | Through the study completion, an average of around 2 years
  Disease Control Rate (DCR) assessed by investigator per RECIST version 1.1
Part A: To assess the anti-tumor activity | Through the study completion, an average of around 2 years
  Percentage change in tumor size assessed by investigator per RECIST version 1.1
Part A: To assess the anti-tumor activity | Through the study completion, an average of around 2 years
  Progression Free Survival (PFS) assessed by investigator per RECIST version 1.1
Part A: To characterize the Pharmacokinetics of DZD6008 | Through the study until the time specified in the protocol, an average of around half year.
  To characterize the concentration of DZD6008 in plasma and cerebrospinal fluid (selected participants with brain metastasis).
Part A: To characterize the Pharmacokinetics of sunvozertinib and DZ0753 | Through the study until the time specified in the protocol, an average of around half year.
  To characterize the concentrations of sunvozertinib and DZ0753 in plasma and cerebrospinal fluid (selected participants with brain metastasis).
Part B: To assess the anti-tumor activity | Through the study completion, an average of around 2 years
  DoR assessed by investigator per RECIST version 1.1
Part B: To assess the anti-tumor activity | Through the study completion, an average of around 2 years
  DCR assessed by investigator per RECIST version 1.1
Part B: To assess the anti-tumor activity | Through the study completion, an average of around 2 years
  Percentage change in tumor size assessed by investigator per RECIST version 1.1
Part B: To assess the anti-tumor activity | Through the study completion, an average of around 2 years
  PFS assessed by investigator per RECIST version 1.1
Part B: To assess safety and tolerability | Through the study completion, an average of around 2 years
  Number of participants with AEs /SAEs
Part B: To characterize the Pharmacokinetics of DZD6008 | Through the study until the time specified in the protocol, an average of around half year.
  To characterize the concentration of DZD6008 in plasma and cerebrospinal fluid (selected participants with brain metastasis).
Part B: To characterize the Pharmacokinetics of sunvozertinib and DZ0753 | Through the study until the time specified in the protocol, an average of around half year.
  To characterize the concentration of sunvozertinib and DZ0753 in plasma and cerebrospinal fluid (selected participants with brain metastasis).

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Beijing Chest Hospital, Beijing, Beijing Municipality
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Zhejiang Taizhou Hospital, Taizhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No